CLINICAL TRIAL: NCT02219386
Title: Dry Needling of the Trapezius Muscle in Office Workers With Neck Pain. Randomised, Single Blinded Clinical Trial
Brief Title: Dry Needling of the Trapezius Muscle in Office Workers With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Ester Cerezo-Téllez, Physical Therapist.Master., University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44/11Comision of investigation
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Myofascial Trigger Point Pain
Keywords: Myofascial pain syndromes,physiotherapy,muscle stretching exercises,neck pain,dry needling
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep dry needling (Active Comparator): The group of DDN receive this treatment and stretch
  Interventions: Other: Group 1. Deep dry needling
- muscle stretch (Other): The stretch applied was as described by Simons et al. (Simons et al., 1999). During the stretch the physiotherapist took up the slack, avoiding pain elicitation, maintaining the tension for four seconds and releasing the tension for eight seconds; this cycle was repeated three times
  Interventions: Other: Group 1. Deep dry needling; Other: group 2. Passive analitical stretch (performed in both groups)

INTERVENTIONS:
Other: Group 1. Deep dry needling — Deep dry needling and stretch. The intervention included DDN of every active MTrP found in the trapezius muscle using a 4 cm x 0.32 mm acupuncture needle as described by Simons et al. (Simons et al., 1999). Once the needle was inserted into the MTrP previously marked by the blinded assessor, local twitch responses (LTRs) were obtained by using Hong's fast-in and fast-out technique, which involves rapid movements of the needle in and out of the MTrP. After four LTRs, the needle was withdrawn and the area was disinfected with alcohol again (Simons et al., 1999). Then, passive stretch was performed on the trapezius muscle.
Other: group 2. Passive analitical stretch (performed in both groups)
  Other Names: only the same stretch as performed in deep dry needling group.
  Arms: muscle stretch

SUMMARY:
Deep dry needling of active myofascial trigger points of trapezius muscle is effective in the dimminution of pain of patients

DETAILED DESCRIPTION:
EVALUATION:

A blind assesor does a complete evaluation of the patients to determine if they take part of the study. An assesment of pain (by visual analogue scale), Pain pressure theshold (kg/cm2 by algometry, Range of motion (CROM goniometer in degrees) and strength (digital dinamometry in Newtons) are performed. In this evaluation inclusion criteria is checked too.

INTERVENTION:

-TREATMENT GROUP(Deep dry needling group (DDN)):

An experienced physical therapist performed this treatment. The intervention included DDN of every active MTrP found in the trapezius muscle using a 4 cm x 0.32 mm acupuncture needle with guided tube. ). In the case of upper trapezius active MTrPs, DDN was performed in the prone position. For medium and lower trapezius muscle MTrPs, DDN was performed in a side-lying position as described by Simons et al. (Simons et al., 1999). Once the needle was inserted into the MTrP previously marked by the blinded assessor, local twitch responses (LTRs) were obtained by using Hong's fast-in and fast-out technique, which involves rapid movements of the needle in and out of the MTrP.

After that, the stretch is performed

- Passive stretch of the trapezius muscle (both groups)

Another experienced physical therapist, after taking part of training-sesions to do the same stretch as in DDN group, performed the stretch.Participants in this group received the same stretch as patients in treatment group.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* present myofascial trigger points in trapezius muscle

Exclusion Criteria:

* to be under anti-inflammatory, analgesic, anticoagulant, muscle relaxant or antidepressant medication at the start of the study or one week before it (Simons, 2004)
* to suffer from fibromyalgia syndrome, or to have any contraindication to conservative or invasive physiotherapy (infection, fever, hypothyroidism, fear of needles, wounds in the area of the puncture, metal allergy, cancer, systemic disease) (Baldry, 2005).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Subjective Pain scored by Visual Analogue Scale (VAS.Participants were followed for the duration of the intervention, an average of 6 weeks) | pretreatment, postreatment and follow-up(15 days)
  pretreatment = at baseline; post-treatment= after 5 physical therapy sessions, 3 weeks after baseline; follow-up= 15 days after last intervention.

SECONDARY OUTCOMES:
Pain Pressure Threshold (PPT. Participants were followed for the duration of the intervention, an average of 6 weeks) | Pretreatment, post treatment and follow-up.
  pretreatment = at baseline; post-treatment= after 5 physical therapy sessions, 3 weeks after baseline; follow-up= 15 days after last intervention.

OTHER OUTCOMES:
Strenght scored by Digital dynamometer (Participants were followed for the duration of the intervention, an average of 6 weeks) | Pretreatment, post treatment and follow-up.
  pretreatment = at baseline; post-treatment= after 5 physical therapy sessions, 3 weeks after baseline; follow-up= 15 days after last intervention.
Cervical Range of Motion assesed with CROM goniometer (Participants were followed for the duration of the intervention, an average of 6 weeks) | Pretreatment, post treatment and follow-up.
  pretreatment = at baseline; post-treatment= after 5 physical therapy sessions, 3 weeks after baseline; follow-up= 15 days after last intervention. Participants were followed for the duration of the intervention, an average of 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ester Cerezo-Téllez, PT, Principal Investigator — Alcalá University
Locations (1):
- UDAIF, Alcalá de Henares, Madrid, Spain